CLINICAL TRIAL: NCT06542848
Title: The Effect of Physiotherapy Rehabilitation Program on Spasticity Level, Upper Extremity Functions, Activities of Daily Living, and Kinesiophobia in Hemiplegic Patients
Brief Title: Impact of Physiotherapy on Spasticity, Upper Limb Function, Daily Activities, and Kinesiophobia in Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Assistant Professor, University of Beykent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBeykent-7
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hemiplegia; Stroke
MeSH Terms: conditions — Hemiplegia; Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): This group consists of patients with post-stroke hemiplegia who will undergo a physiotherapy and rehabilitation program to assess its effects on spasticity levels, upper extremity functions, activities of daily living, and kinesiophobia.
  Interventions: Other: Physiotherapy and Rehabilitation Practices

INTERVENTIONS:
Other: Physiotherapy and Rehabilitation Practices — The treatment program consisted of 3 sessions per week, each lasting 45 minutes. The rehabilitation program included 30 minutes of conventional TENS application to the wrist extensor muscles and quadriceps muscle, upper and lower extremity exercises, balance and coordination exercises, and weight transfer exercises. The upper extremity exercises consisted of range of motion exercises for the shoulder joint, while the lower extremity exercises included range of motion exercises for the hip, knee, and ankle joints. Balance exercises included forward, backward, and lateral leaning exercises, as well as weight transfer and stepping exercises in all directions. The treatment duration was planned to be a total of 24 sessions over 8 weeks. Evaluations were conducted before and after the treatment program.

SUMMARY:
This study investigated the effects of rehabilitation exercises on spasticity levels, upper extremity functions, activities of daily living, and kinesiophobia in patients with hemiplegia following a stroke.

DETAILED DESCRIPTION:
Hemiplegia is a neurological condition characterized by paresis and movement limitations on one side of the body due to functional loss in one hemisphere of the brain caused by a vascular event after a stroke. This study aims to evaluate the effects of a physiotherapy and rehabilitation program on spasticity levels, upper extremity functions, activities of daily living, and kinesiophobia in patients with post-stroke hemiplegia.

Participants' spasticity levels were assessed using the Modified Ashworth Scale, upper extremity functions with the Fugl-Meyer Upper Extremity Motor Assessment, activities of daily living with the Barthel Index, and kinesiophobia levels with the Tampa Scale of Kinesiophobia. The treatment program consisted of 24 sessions, with three sessions per week. Each session lasted 45 minutes and included Transcutaneous Electrical Nerve Stimulation (TENS), range of motion exercises for upper and lower extremities, balance and coordination exercises, and weight transfer exercises. Assessments were conducted before and after the treatment.

As a result of the treatment program, a significant decrease in spasticity levels was observed in joints other than the hip joint, along with significant improvements in upper extremity functions and activities of daily living, and a significant reduction in kinesiophobia levels.

Physiotherapy and rehabilitation programs have been found to be effective in reducing spasticity, improving upper extremity functions and activities of daily living, and reducing kinesiophobia in post-stroke hemiplegic patients. These findings can contribute to the development of post-stroke rehabilitation strategies. Future research should deepen these findings with larger sample groups and long-term follow-up studies.

ELIGIBILITY:
Inclusion Criteria:

* Being between 22-79 years of age
* Having been diagnosed with a stroke (SVO)
* Possessing adequate language and cognitive skills
* Willingness to participate voluntarily
* Not having any chronic diseases that could affect the study outcomes

Exclusion Criteria:

* No other neurological problems affecting functionality besides hemiplegia
* Having cognitive impairment

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Effect of Rehabilitation Program on Spasticity with Modified Ashworth Scale | Baseline (pre-treatment) and 8 weeks (post-treatment)
  The primary outcome measure evaluates the changes in spasticity levels. The Modified Ashworth Scale is a measurement system based on manually assessing the resistance of specific muscle groups to passive movement. This scale evaluates the resistance encountered during passive movement of the extremity, scoring it from 0 to 4. As the score increases, it indicates a higher level of spasticity.
Effect of Rehabilitation Program on Upper Extremity Motor Function with Fugl-Meyer Assessment of Upper Extremity Motor Function | Baseline (pre-treatment) and 8 weeks (post-treatment)
  The Fugl-Meyer Assessment of Upper Extremity Motor Function is a disease-specific, objective motor impairment scale designed to evaluate recovery in hemiplegic patients following a stroke. The highest possible score on this assessment is 66. An increase in the score indicates better motor skills.
Effect of Rehabilitation Program on Daily Living Activities with Barthel Index of Activities of Daily Living | Baseline (pre-treatment) and 8 weeks (post-treatment)
  The Barthel Index of Activities of Daily Living consists of 10 items related to daily activities and mobility. The highest possible total score is 100, indicating that the individual is completely independent in their physical functions. The lowest score is 0, indicating that the individual is entirely dependent.
Effect of Rehabilitation Program on Kinesiophobia with Tampa Scale for Kinesiophobia | Baseline (pre-treatment) and 8 weeks (post-treatment)
  The Tampa Scale for Kinesiophobia is a self-report measure developed to assess fear of movement. It consists of 17 items. A high score indicates a high level of fear of movement, while a low score indicates a negligible level of fear of movement. The total score, obtained by summing the individual items, ranges from 17 to 68.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, PhD, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No